CLINICAL TRIAL: NCT00140452
Title: Phase II Study Using Thalidomide for the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: Phase II Study Using Thalidomide for the Treatment of ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Celgene Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALS-001
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2007-11-21 (Estimated); Status verified 2007-11

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Thalidomide — Thalidomide will start at a dose of 100mg/day, dose escalated every 2 weeks by 100mg/day to a target dose of 400mg/day.

SUMMARY:
The use of Thalidomide in patients with ALS who have disease progression.

DETAILED DESCRIPTION:
Phase II open labeled trial testing the efficacy of thalidomide for ALS in the setting of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Clinically proven ALS
* Disease duration less than or equal to 5 years
* ALSFRS-R score equal to or greater then 30

Exclusion Criteria:

* Patients with known deep venous thrombosis or hyper coagulable state will be excluded
* Patients with FVC less than 80%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-02; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of Thalidomide in the rate of progression in ALS at 9 months and hence determine preliminary efficacy in the treatment of ALS | Efficacy will be gauged according to the slopeof the expected average decline at nine months after starting Thalidomide

SECONDARY OUTCOMES:
To evaluate 1) toxicity 2) quality of life 3) cytokine profile 4) PFT's 5) sleep questionnaire and 6) survival of thalidomide in the treatment of ALS | survival and progression free suvival will be assessed from the date of initial therapy on study to date od death. Survival and progresion free survival wil be analyzed using the Kaplan Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Elijah Stommel, Principal Investigator
Locations (1):
- Dartmouth Hichcock Medical Center, Lebanon, New Hampshire, United States